CLINICAL TRIAL: NCT02537106
Title: A Comparison of the Effect of 1.5% Versus 3% NaCl on Brain Relaxation and Microcirculation During the Supratentorial Brain Tumor Surgery, and Natremia and Osmolarity in Postoperative Period
Brief Title: A Comparison of the Effect of 1.5 Versus 3% NaCl on Brain Relaxation and Microcirculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Dostalova Vlasta, MD, PhD, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201508-S23P
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Brain Tumors
Keywords: Brain Tumors; Microcirculation; Osmotherapy; Hypertonic NaCl; Natremia
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.5% NaCl (Experimental): After standardized induction to general anesthesia group A patients will be given the infusion of hyperosmotic 1.5% NaCl 5 ml/kg/BW during 15 min.
  Interventions: Procedure: 1.5% NaCl
- 3% NaCl (Experimental): After standardized induction to general anesthesia group B patients will be given the infusion of hyperosmotic 3% NaCl 5 ml/kg/BW during 15 min.
  Interventions: Procedure: 3% NaCl

INTERVENTIONS:
Procedure: 1.5% NaCl — After the infusion of 1.5% NaCl and dura opening the microcirculation and the brain relaxation score will be measured in the area of healthy brain and perifocal oedema sites. Microcirculation measurement will be repeated at the same sites after tumor resection.
  Arms: 1.5% NaCl
Procedure: 3% NaCl — After the infusion of 3% NaCl and dura opening the microcirculation and the brain relaxation score will be measured in the area of healthy brain and perifocal oedema sites. Microcirculation measurement will be repeated at the same sites after tumor resection.
  Arms: 3% NaCl

SUMMARY:
Hyperosmotic solutions of 1.5% and 3% NaCl are equally effective for brain relaxation and microcirculation during brain surgery. The effect of 1.5% NaCl on postoperative natremia and natriuresis is less pronounced.

DETAILED DESCRIPTION:
All the patients meeting the study criteria will be randomized into two groups. After standardized induction to general anesthesia all patients will be given the infusion of hyperosmotic NaCl 5 ml/kg/BW during 30 min, group A 1.5% NaCl, group B 3% NaCl. Corticosteroids will be administered as usually. After dura opening the brain relaxation score will be assessed by surgeon (1 = completely relaxed, 2 = satisfactorily relaxed, 3 = firm brain, 4 = bulging brain), and the first measurement of the brain microcirculation provided by use of SDF probe in the area of the healthy brain, and of perifocal oedema. Both sites of investigation will be marked for the second measurement, which will be done after the end of tumor resection. Laboratory examinations: natremia preoperatively, natremia and osmolarity peroperatively 1 hour after NaCl infusion and at the end of surgery. Concentration of natrium will be examined in CSF after dura opening. Anesthesia management will be according to the standardised protocol, the patients will be awaken and extubated after the end of the procedure at the operating theatre.

ELIGIBILITY:
Inclusion Criteria:

* peripheral supratentorial brain tumors or metastasis
* indication for osmotherapy
* ASA status I-III

Exclusion Criteria:

* reoperation
* osmotherapy prior to surgery
* preoperative natremia less than 135 mmol/l and more than 140 mmol/l
* GCS less than 14
* obstructive hydrocephalus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Changes in brain microcirculation | from dura opening till the end of tumor resection
  measurement by SDF probe MicroVision

SECONDARY OUTCOMES:
Changes in natremia | 1 hour after hypertonic NaCl infusion
  mmol/l
Changes in natremia | 5 min after the end of surgery
  mmol/l
Changes in osmolarity | 1 hour after hypertonic NaCl infusion
  mosm/l
Changes in osmolarity | 5 min after the end of surgery
  mosm/l
Concentration of natrium in cerebrospinal fluid | after dura opening
  mmol/l

OTHER OUTCOMES:
Changes in diuresis | at the time of extubation
  ml/hour

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Dostalova, MD., Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia